CLINICAL TRIAL: NCT02964585
Title: Role of Canagliflozin on Gene Expression and Function of CD34+ Endothelial Progenitor Cells and Renal Function in Patients With Type 2 Diabetes
Brief Title: Role of Canagliflozin on CD34+ Cells in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Sabyasachi Sen, Associate Professor of Medicine, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GW-CANA-081635
Record Dates: First submitted 2016-10-06; First posted 2016-11-16 (Estimated); Results first posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Endothelial Cells; Cellular Biomarker; Endothelial Dysfunction; CD34+; Impaired renal function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Arm (Active Comparator): 100 mg of Canagliflozin for 16 weeks
  Interventions: Drug: Canagliflozin
- Placebo Arm (Placebo Comparator): Placebo for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin — 100 mg
  Other Names: INVOKANA
  Arms: Active Arm
Drug: Placebo — 1 tablet daily for 16 weeks
  Arms: Placebo Arm

SUMMARY:
The investigators hypothesize that Cana may be able to improve number and function of CD34+ endothelial progenitor cells. The investigators also propose that this expected cardiovascular benefit is independent of HbA1C reduction.

Subjects will begin taking 100 mg of Cana or placebo after initial 4 weeks. Subjects will be withdrawn from the study if the medication or placebo is not tolerated.

DETAILED DESCRIPTION:
Diabetes affects more than 11% of adults in the United States and this is projected to nearly double by 2025. Both diabetes and obesity are associated with endothelial dysfunction, oxidative stress, endothelial cell inflammation, cardiovascular pro-thrombotic states and are the most common causes of kidney disease. Use of a sodium-glucose linked transporter (SGLT-2) inhibitor has shown promise in improving glycemic control, weight reduction, hypertension and even changes in circulating Renin-angiotensin-aldosterone system (RAAS) and nitric oxide (NO). However, whether these group of drugs have any effect on cardiovascular disease (CVD) risk modification or on endothelium or endothelial progenitor cells as a surrogate of cardiovascular and renal risk outcome measure, is unclear.

The investigators have previously shown that CD34+ cells, derived from peripheral blood can act as a cellular biomarker that is more reliable than serum based markers for CVD risk estimation. Serum based inflammatory markers are not useful until the endothelium is already damaged and inflamed. Such serum based biomarkers takes several months to change and gives no preventive and predictable information as to whether a particular medication may affect future endothelium. This is why the study of endothelium progenitors is crucial. In the investigators' previous study of a prediabetes population with an aerobic exercise intervention, the investigators have demonstrated that CD34+ cells are responsive to a change in therapy or intervention within 2-4 weeks and can be used as a reliable non serum based cellular bio-marker. CD34+ cells or endothelial progenitor cells have been used clinically to improve collateral circulation and have been extensively studied as a robust cardiovascular biomarker. Therefore studying CD34+ cells in patients, with or without Canagliflozin (Cana) can give vital information about the medication and its effect on endothelium. This is particularly important as another SGLT2 inhibitor Empagliflozin has shown unparalleled positive cardiovascular effects with an oral hypoglycemic agent. Of course, the question arises whether this clinical trial effect is secondary to glucose effect or direct effect of SGLT2 inhibitor on endothelium.

Multiple glucose transporters have been identified in human cells these include GLUTs, SGLTs and even taste receptors (such as TLR2 and TLR3). The investigators know SGLT transporters are present in tubular cells and clearly blocking of SGLT2 in these cells is beneficial. Information on glucose transporter in stem or progenitor cells is almost nil. In our lab the investigators have shown presence of GLUT1, SGLTs and TLR3 on CD34+ cells. The investigators have also demonstrated that hyperglycemia is toxic to CD34+ cells, more than CD31+ positive mature endothelial cells. The investigators hypothesize that blocking SGLT2 in CD34+ cells will be beneficial rather than detrimental. As far as glucose uptake in CD34+ cells are concerned other glucose transporters should be sufficient, in fact lesser amount of glucose entry in a hyperglycemic milieu (type 2 DM patients) may be less pro-inflammatory and less pro-apoptotic.

Our preliminary data indicates that mRNA gene expression of both SGLT1 and SGLT2 are noted on human CD34+ cells however only SGLT2 mRNA gene expression is up-regulated several fold in human CD34+ cells in presence of hyperglycemia (20mM glucose). However non primary commercially obtained human endothelium (HUVEC) do not show similar results. An explanation could be SGLT2 expression decreases as the cell transitions from progenitor to mature endothelium. From these results the investigators believe SGLT2 inhibitor will be effective on progenitors and not mature endothelium. The investigators therefore hypothesize that CD34+ cells will be an ideal biomarker to study the effect of the drug. It is possible that Cana, by blocking SGLT2 receptors, may influence other CD34+ cell surface receptors including other glucose transporters and influence its function (most importantly migration). If a particular medication positively influences stem/progenitor cell migration then that medication can positively influence endothelial dysfunction and vascular complications from diabetes. The investigators are particularly interested to note effect of Canagliflozin, a SGLT2 inhibitor on other glucose transporters such as GLUT 1 and 4 while looking at SGLT 1 and 2 on CD34+ cells. It will be helpful to discern these effects particularly when choice of oral diabetic medication in a type 2 diabetes population is practically limited to metformin, DPP4 inhibitors and SGLT2 inhibitors. The investigators plan to investigate the effect of Cana on CD34+ cells, in a placebo matched study. The investigators plan to recruit subjects with type 2 diabetes with the following characteristics: 1) overweight, mild and moderately obese (BMI=25.0-39.9); 2) individuals with early type 2 diabetes (≤15 years) with inadequate control, HbA1C= 7.0 to 10.0%, on Metformin (1-2 grams/day) 3) with no history or presence of macrovascular complication and CKD no higher than stage 2. The subjects will be on Metformin as per ADA, Metformin is the 1st line of care along with life-style modification. While Metformin on its own may affect inflammatory biomarkers, the effect is minimal at best, particularly in presence of CKD and endothelial dysfunction. Also both placebo and the cana group will be on Metformin.

The investigators will recruit a total of 40 patients (20 individuals/per group) with approximately a 20% drop out rate over two years and the investigators hope to retain 32 individuals (16/group). Individuals in each group will be matched by sex, age, and race. Participants will be assessed at baseline (week 0), and at 2 and 4 months of drug intake.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-70 years
* Currently treated with any combination of the following anti-diabetic therapies: metformin (1-2 grams), insulin, GLP-1 agonists, a DPP-IV inhibitor, or sulfonylureas
* Hemoglobin A1C (HbA1C) between 7.0% and 10.0%
* Body Mass Index (BMI) between 25 and 39.9 kg/m^2 (both inclusive)

Exclusion Criteria:

* Type 1 diabetes
* History of hyperosmolar nonketotic coma
* History of diabetic ketoacidosis in the last 3 months
* Abnormal CBC that is judged by physician to be unsafe to enroll or low hematocrit (<28 UNITS).
* History of pancreatitis
* History of diabetic ketoacidosis in the last 3 months
* History of cancer (except basal cell carcinoma and cancer that is cured or not active or being treated in the past 5 years)
* Heart attack or stroke within 6 months of screening
* Clinically significant coronary and/or peripheral vascular disease that would be unsafe to enroll in the study.
* Statin use started or dose change in the last 3 months
* CKD Stages 3,4 and 5
* Use of oral or injectable anti-diabetic medication other than any combination of the following anti-diabetic therapies: metformin (1-2 grams), insulin, GLP-1 agonists, a DPP-IV inhibitor, or sulfonylureas currently, or in the past 1 month.
* Use of consistent long-term steroid medication (oral, inhaled, injected) within the last 3 months
* Uncontrolled inflammatory disease, or current chronic use of anti-inflammatory drugs within the last 3 months. **This will be judged on a case by case basis by the PI**
* Implanted devices (e.g., pacemakers) that may interact with Body Composition scale
* Untreated Systolic Blood Pressure > 150 mmHg and diastolic Blood Pressure > 90 mmHg
* Active wounds or recent surgery within 3 months
* Untreated hyper/hypothyroidism

Physical and Laboratory Test Findings:

* Pre-existing liver disease and/or ALT and AST >2.5X's UNL
* Serum creatinine levels ≥2.0
* Estimated CrCl < 60 mL/min (measured by eGFR value)
* Triglycerides >450 mg/dL

Allergies and Adverse Drug Reactions:

* Subjects with a history of any serious hypersensitivity reaction to Cana or another SGLT2 inhibitor.

Sex and Reproductive Status:

* Women in reproductive age group will be included in the study but encouraged to use contraceptive method to avoid pregnancy within 16 weeks of study duration.
* Women who are pregnant or breast-feeding will be excluded.

Other Exclusion Criteria:

* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
* Patients who are active smokers
* Patients who are pregnant
* Nursing women
* Post-menopausal women who are on estrogen hormone replacement therapy will be excluded.
* Patients on low dose oral contraceptives will be allowed to participate as these formulations contain very low amounts of estrogens.
* Eligibility criteria for this study have been carefully considered to ensure the safety of the study subjects and to ensure that the results of the study can be used. It is imperative that subjects fully meet all eligibility criteria.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabyasachi Sen, MD, PhD, Principal Investigator — Medical Faculty Associates
Locations (1):
- The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sen S, Strappe PM, O'Brien T. Gene transfer in endothelial dysfunction and hypertension. Methods Mol Med. 2005;108:299-314. doi: 10.1385/1-59259-850-1:299. PMID 16028691
- [Background] Krenning G, Dankers PY, Drouven JW, Waanders F, Franssen CF, van Luyn MJ, Harmsen MC, Popa ER. Endothelial progenitor cell dysfunction in patients with progressive chronic kidney disease. Am J Physiol Renal Physiol. 2009 Jun;296(6):F1314-22. doi: 10.1152/ajprenal.90755.2008. Epub 2009 Apr 1. PMID 19339628
- [Background] Department of Health and Human Services, NIH and National Center for Chronic Disease Prevention and Health Promotion, "National Diabetes Statistics: 2007 and 2011 Fact Sheet." 2011
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] Afkarian M, Sachs MC, Kestenbaum B, Hirsch IB, Tuttle KR, Himmelfarb J, de Boer IH. Kidney disease and increased mortality risk in type 2 diabetes. J Am Soc Nephrol. 2013 Feb;24(2):302-8. doi: 10.1681/ASN.2012070718. Epub 2013 Jan 29. PMID 23362314
- [Background] Rask-Madsen C, King GL. Mechanisms of Disease: endothelial dysfunction in insulin resistance and diabetes. Nat Clin Pract Endocrinol Metab. 2007 Jan;3(1):46-56. doi: 10.1038/ncpendmet0366. PMID 17179929
- [Background] Stanton RC. Sodium glucose transport 2 (SGLT2) inhibition decreases glomerular hyperfiltration: is there a role for SGLT2 inhibitors in diabetic kidney disease? Circulation. 2014 Feb 4;129(5):542-4. doi: 10.1161/CIRCULATIONAHA.113.007071. Epub 2013 Dec 13. No abstract available. PMID 24334174
- [Background] Oliva RV, Bakris GL. Blood pressure effects of sodium-glucose co-transport 2 (SGLT2) inhibitors. J Am Soc Hypertens. 2014 May;8(5):330-9. doi: 10.1016/j.jash.2014.02.003. Epub 2014 Feb 12. PMID 24631482
- [Background] Sabyasachi Sen, Sarah Witkowski, Ann Lagoy, Ashequl M. Islam: A six-week home exercise program improves endothelial function and CD34+ circulating progenitor cells in patients with pre-diabetes. J Endocrinol Metab.2015; 5 (1-2):163-171, doi: http://dx.doi.org/10.14740/jem273w.
- [Background] Werner N, Kosiol S, Schiegl T, Ahlers P, Walenta K, Link A, Bohm M, Nickenig G. Circulating endothelial progenitor cells and cardiovascular outcomes. N Engl J Med. 2005 Sep 8;353(10):999-1007. doi: 10.1056/NEJMoa043814. PMID 16148285
- [Background] Losordo DW, Schatz RA, White CJ, Udelson JE, Veereshwarayya V, Durgin M, Poh KK, Weinstein R, Kearney M, Chaudhry M, Burg A, Eaton L, Heyd L, Thorne T, Shturman L, Hoffmeister P, Story K, Zak V, Dowling D, Traverse JH, Olson RE, Flanagan J, Sodano D, Murayama T, Kawamoto A, Kusano KF, Wollins J, Welt F, Shah P, Soukas P, Asahara T, Henry TD. Intramyocardial transplantation of autologous CD34+ stem cells for intractable angina: a phase I/IIa double-blind, randomized controlled trial. Circulation. 2007 Jun 26;115(25):3165-72. doi: 10.1161/CIRCULATIONAHA.106.687376. Epub 2007 Jun 11. PMID 17562958
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Result] Nandula SR, Kundu N, Awal HB, Brichacek B, Fakhri M, Aimalla N, Elzarki A, Amdur RL, Sen S. Role of Canagliflozin on function of CD34+ve endothelial progenitor cells (EPC) in patients with type 2 diabetes. Cardiovasc Diabetol. 2021 Feb 13;20(1):44. doi: 10.1186/s12933-021-01235-4. PMID 33581737

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Arm | Placebo Arm
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm | Placebo Arm | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.64 (7.75) | 59.15 (11.24) | 57.72 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.71 (1.41) | 33.11 (1.08) | 31.55 (0.92)
Body Fat Percentage [Mean (Standard Deviation); unit: percentage of body fat] | 32.92 (2.39) | 39.65 (2.64) | 36.14 (1.86)
HbA1C [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.39 (0.36) | 7.93 (0.33) | 8.14 (0.24)
eGFR [Mean (Standard Deviation); unit: mL/min] | 80.24 (4.27) | 85.22 (4.43) | 82.43 (3.08)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.96 (0.05) | 0.84 (0.05) | 0.90 (0.04)
HDL [Mean (Standard Deviation); unit: mg/dL] | 42.96 (3.47) | 51.56 (3.60) | 47.0 (2.50)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 167.78 (9.74) | 163.40 (10.09) | 166.60 (7.08)
LDL/HDL [Mean (Standard Deviation); unit: unitless (ratio)] | 2.19 (0.15) | 1.68 (0.15) | 1.94 (0.13)
C-reactive Protein [Mean (Standard Deviation); unit: mg/dL] | 0.54 (0.2) | 1.03 (0.2) | 0.79 (0.2)
Insulin [Mean (Standard Deviation); unit: mg/dL] | 2.50 (0.20) | 2.49 (0.21) | 2.50 (0.20)
Augmentation Index [Mean (Standard Deviation); unit: Percent Aug pressure of Pulse Pressure] — Defined as Augmentation Pressure/Pulse Pressure * 100. Higher values generally correspond to increased risk of CVD.
  Percent Aug pressure of Pulse Pressure | 24.2 (2.8) | 22.1 (2.9) | 22.95 (1.94)
Pulse wave velocity [Mean (Standard Deviation); unit: m/s] — calculated via delay of pulse reaching femoral artery versus carotid artery, divided by the difference in distance of each measurement point from the aortic notch
  m/s | 9.59 (0.66) | 11.19 (0.64) | 10.81 (0.40)
Leptin [Mean (Standard Deviation); unit: ug/dL] | 28.36 (3.30) | 39.84 (3.34) | 33.29 (4.02)
SDF-1a [Mean (Standard Deviation); unit: pg/mL] | 5.49 (0.46) | 6.34 (0.47) | 5.92 (0.46)
3-hydroxy-butyric acid [Mean (Standard Deviation); unit: mmol/mol Creatinine] | 0.01 (0.01) | 0.03 (0.01) | 0.01 (0.02)
Acetoacetic Acid [Mean (Standard Deviation); unit: mmol/mol Creatinine] | 1.08 (0.24) | 0.72 (0.25) | 0.90 (0.24)
Mean MNC [Mean (Standard Deviation); unit: cells*10^6/mL] | 147.75 (15.54) | 167.00 (16.08) | 157.04 (10.41)
%CD34+ [Mean (Standard Deviation); unit: percentage of MNCs] | 0.94 (0.19) | 1.01 (0.19) | 0.98 (0.18)
Nephrin [Mean (Standard Deviation); unit: ug/dL] | 5.39 (0.51) | 6.15 (0.55) | 5.77 (0.54)
PODXL [Mean (Standard Deviation); unit: ug/dL] | 7.05 (0.31) | 6.72 (0.33) | 6.89 (0.31)
Colony Forming Units [Mean (Standard Deviation); unit: CFU] — Assesses differentiation and proliferation of stem cells by plating a certain number of cells into a controlled dish, and counting the colonies formed after 14 days.
  CFU | 6.08 (1.95) | 10.30 (2.03) | 8.14 (0.98)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 125.79 (3.07) | 125.77 (5.28) | 125.78 (2.98)
  Diastolic | 81.14 (2.04) | 74.92 (1.94) | 78.34 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: Gene Expression and Function Change of CD34+ Endothelial Progenitor Cells (Protein Expression)
Description: To determine whether 4 months of Canagliflozin modifies CD34+ cell number, gene expression and migration function. The investigators will obtain a total of approximately 95 mL of peripheral blood per visit. Of these 95 mL, 60-70 mL will be used to obtain CD34+ cells from mononuclear cell (MNC) population and 25-35 mL for biochemistry and plasma ELISA assays. MNC will be obtained from whole blood similar to protocols described before [13,14]. MNCs will be put through CD34 magnetic bead column to obtain CD34+ cells (Miltenyi Biotec). Purity of CD34+ cells, post sort, usually is above 90%, to be verified by FACS analysis.
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Deviation); unit: ng/mL in serum
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
ng/mL in serum
  CXCL12 Expression | 0.63 (0.18) | 0.33 (0.17)
  CXCR4 Expression | 1.58 (0.18) | 0.90 (0.18)
  EDN1 | 2.10 (0.27) | 1.03 (0.29)
  VEGEF-A | 1.12 (0.19) | 0.83 (0.19)
  PECAM | 1.28 (0.12) | 0.89 (0.12)
  KDR | 1.16 (0.2) | 0.5 (0.2)
  NOS3 | 0.34 (0.21) | -0.25 (0.21)
  Catalase | 0.20 (0.26) | -0.61 (0.26)
  GPX35 | 2.25 (0.54) | 1.71 (0.54)
  SDF 10 NG | 0.26 (0.03) | 0.23 (0.03)
  SOD2 | 1.36 (0.24) | 0.92 (0.24)

2. Primary Outcome: Gene Expression and Function Change of CD34+ Endothelial Progenitor Cells (Cell Percentages)
Description: as for outcome 1
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Deviation); unit: percentage of MNCs
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
percentage of MNCs
  Percent of CD34+ | 0.93 (0.17) | 1.23 (0.21)
  Percent of CD31+ | 2.58 (0.35) | 2.16 (0.43)
  Percent CD34+ and CD184+ | 0.37 (0.09) | 0.61 (0.11)

3. Primary Outcome: Gene Expression and Function Change of CD34+ Endothelial Progenitor Cells (Cell Counts)
Description: as for outcome 1
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Deviation); unit: cells*10^6/mL
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
cells*10^6/mL
  Mean MNC count | 155.09 (15.54) | 155.09 (16.08)
  Mean CD34+ve cell count (x100) | 2682.93 (491.44) | 3157.36 (508.69)

4. Primary Outcome: Gene Expression and Function Change of CD34+ Endothelial Progenitor Cells (Cell Proliferation)
Description: as for outcome 1
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Deviation); unit: Colony forming units (CFU)
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
Colony forming units (CFU) | 7.53 (1.89) | 13.69 (2.10)

5. Secondary Outcome: Serum Endothelial Inflammatory Markers (1)
Description: IL-6, and TNF-alpha
Time Frame: measured at 8 and 16 (reported) weeks post treatment
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-6 | 4.56 (4.91) | 3.21 (1.82)
  TNF-alpha | 1.36 (0.34) | 1.63 (0.53)

6. Secondary Outcome: Fasting Lipid Profile
Description: Measured from a serum blood Lipid Panel: cholesterol and serum ketone bodies
Time Frame: 16 weeks post Canagliflozin treatment reported (also measured at 8 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
mg/dL
  Cholesterol | 171.57 (9.84) | 147.76 (10.61)
  HDL | 46.17 (3.48) | 51.67 (3.69)
  LDL | 96.03 (6.93) | 82.672 (8.27)
  3-hydroxybutyric acid (ketone body) | 0.02 (0.01) | 0.03 (0.01)
  Acetoacetic acid (ketone body) | 0.69 (0.24) | 0.30 (0.27)

7. Secondary Outcome: Glycemic Control (HbA1C)
Description: As determined by HbA1C values
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
percentage of hemoglobin | 7.85 (1.66) | 8.26 (1.52)

8. Secondary Outcome: BMI
Description: Determined as weight in kg divided by height in meters squared
Time Frame: 16 weeks post Canagliflozin treatment
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
kg/m^2 | 30.53 (1.29) | 34.64 (1.36)

9. Secondary Outcome: Resting Metabolic Rate (RMR)
Description: Using ReeVue (trademark) machine, with or without SGLT2 inhibitor therapy to ascertain if Cana has any effect on RMR. Other related trials have shown weight loss but effect on metabolic rate has not been studied .
Time Frame: 16 weeks post Canagliflozin treatment
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
kcal/day | 1999.31 (67.45) | 1863.01 (165.91)

10. Secondary Outcome: Pulse Wave Velocity
Description: Vessel health assessed by using arterial tonometry with the SphygmoCor CP system from ATCOR .
Time Frame: 16 weeks post Canagliflozin treatment reported (also measured at 8 weeks)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
m/s | 10.12 (0.63) | 11.42 (0.70)

11. Secondary Outcome: Serum Endothelial Inflammatory Markers (2)
Description: Highly selective C-reactive protein (hs-CRP)
Time Frame: measured at 8 and 16 (reported) weeks post treatment
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
mg/L | 0.63 (0.2) | 0.92 (0.2)

12. Secondary Outcome: Glycemic Control
Description: Measured from blood glucose values (fasting) during visit
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
mg/dL | 142.79 (45.24) | 158.0 (38.4)

13. Secondary Outcome: Body Fat Percentage
Description: Measured using a Tanita body composition scale
Time Frame: 16 weeks post Canagliflozin treatment
Measure: Mean (Standard Error); unit: percentage of body mass
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
percentage of body mass | 32.46 (2.32) | 38.58 (2.63)

14. Secondary Outcome: Augmentation Index (Pulse Wave Analysis)
Description: Vessel health assessed by using arterial tonometry with the SphygmoCor CP system from ATCOR. Higher values generally correlate with increased cardiovascular risk.
Time Frame: 16 weeks post Canagliflozin treatment reported (also measured at 8 weeks)
Measure: Mean (Standard Deviation); unit: percent aug pressure of pulse pressure
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
percent aug pressure of pulse pressure | 28.67 (2.8) | 21.37 (3.2)

15. Secondary Outcome: Kidney Function Markers
Description: Creatinine Clearance and Kidney Function measured from compiled results from a urine sample and blood tests
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Error); unit: ug/dL
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
ug/dL
  PODXL | 6.62 (0.30) | 6.68 (0.4)
  Nephrin | 5.24 (0.50) | 5.87 (0.65)
  Wilm's Tumor | 5.75 (0.59) | 6.36 (0.75)

16. Secondary Outcome: Creatinine (Urine)
Description: Creatinine Clearance and Kidney Function measured from compiled results from a urine sample and blood tests
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
mmol/L | 77.08 (15.58) | 106.23 (15.62)

17. Secondary Outcome: Microalbumin
Description: Creatinine Clearance and Kidney Function measured from compiled results from a urine sample and blood tests
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Error); unit: mg/g creatinine
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
mg/g creatinine | 33.97 (13.24) | 43.41 (26.17)

18. Secondary Outcome: eGFR
Description: Creatinine Clearance and Kidney Function measured from compiled results from a urine sample and blood tests
Time Frame: 16 weeks post Canagliflozin treatment reported
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 15 | 14
mL/min | 79.90 (4.21) | 88.33 (4.52)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from signing of consent form to 30 days after last treatment day, approximately 20 weeks in total.
Arm/Group | Active Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

LIMITATIONS AND CAVEATS:
Limitations of our pilot study may include the relatively short 16-week Canagliflozin therapy, which may be inadequate to see significant changes in certain clinical and cellular parameters. This maybe also because of the small sample size. Further studies with a larger population and longer duration may be helpful to further define the mechanisms behind our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT02964585/Prot_SAP_000.pdf